CLINICAL TRIAL: NCT06573294
Title: A First-In-Human, Open-Label, Dose Escalation Trial to Evaluate the Safety and Antitumor Activity of GEN1057 in Subjects With Malignant Solid Tumors
Brief Title: Trial to Assess the Safety and Antitumor Activity of GEN1057 in Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCT1057-01; 2024-513563-75-00 (EU CTIS Number); jRCT2031240508 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-08-26; First posted 2024-08-27 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Advanced Malignant Solid Tumors; Metastatic Malignant Solid Tumors
MeSH Terms: interventions — Premedication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GEN1057 Monotherapy (Experimental)
  Interventions: Drug: GEN1057; Drug: Premedication

INTERVENTIONS:
Drug: GEN1057 — Intravenous (IV) infusion
Drug: Premedication — IV infusion/orally by mouth.

SUMMARY:
The purpose of this trial is to study the antibody GEN1057 when used as a single agent for the treatment of certain types of cancer.

Trial details include:

* The trial duration for an individual participant will be up to approximately 11 months.
* The treatment duration for an individual participant will be up to approximately 4 months (the duration of treatment may vary for each participant) and the follow-up duration for an individual participant will be approximately 6 months.

Participation in the trial will require visits to the site. All participants will receive active drug; no one will be given placebo.

DETAILED DESCRIPTION:
The trial is a first-in-human (FIH) open-label, multicenter, multinational safety trial.

The dose escalation will evaluate different dose levels by assessing safety, tolerability, and early efficacy signals to determine the expansion dose(s) of GEN1057 as monotherapy, as well as characterizing the pharmacokinetic (PK) profile and immunogenicity in participants with malignant solid tumors who have metastatic or advanced disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Advanced and/or metastatic malignant solid tumors, who have progressed on standard of care therapy for whom there is no available standard therapy likely to provide clinical benefit, or who are not candidates for available therapy, and for whom experimental therapy with GEN1057 may be beneficial, in the opinion of the investigator.
* Be at least 18 (or the legal age of consent in the jurisdiction in which the trial is taking place) years of age.
* Have measurable disease according to RECIST v1.1.
* Have Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 1 at screening and on C1D1 pretreatment. Note: If screening ECOG PS is assessed within 3 days prior to C1D1, ECOG PS does not need to be reassessed at C1D1.
* Have a life expectancy of ≥3 months.

Key Exclusion Criteria:

* Has been exposed to any of the following prior therapies/treatments within the specified timeframes:

  * Treatment with an investigational anticancer agent within 28 days or for systemic therapies within 5 half-lives of the drug, whichever is shorter, prior to trial treatment administration.
  * Treatment with an investigational drug, including investigational vaccines within 28 days before the planned first dose of trial treatment.
  * Prior treatment with live, attenuated vaccines within 28 days prior to initiation of GEN1057. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live, attenuated vaccines and are not allowed. Experimental and/or nonauthorized severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccinations are not allowed.
  * Used an invasive investigational medical device within 28 days before the planned first dose of trial treatment.
* Has clinically significant toxicities from previous anticancer therapies that have not resolved to baseline levels or to grade 1, except for anorexia, hyperthyroidism, hypothyroidism, and peripheral neuropathy, which must have recovered to ≤ grade 2. There is no limitation for alopecia and hearing impairment from previous therapies.
* Has known, symptomatic brain metastases. Asymptomatic brain metastases are allowed provided that they have been treated, have been stable for >28 days as documented by radiographic imaging, and do not require prolonged (>14 days) systemic corticosteroid therapy.
* Has a past or current malignancy other than inclusion diagnosis.

Note: Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (AEs) | From first dose until the end of the safety follow-up period (approximately 5 months)
Number of Participants With Dose Limiting Toxicities (DLTs) | Up to 21 days
  DLTs will be graded for severity according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), v5.0.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of GEN1057 | Predose and postdose at multiple timepoints up to end of treatment (approximately 4 months)
Time to Reach Cmax (Tmax) of GEN1057 | Predose and postdose at multiple timepoints up to end of treatment (approximately 4 months)
Area Under the Concentration-time Curve (AUC) From Time Zero to Last Quantifiable Sample (AUC0-last) of GEN1057 | Predose and postdose at multiple timepoints up to end of treatment (approximately 4 months)
Half-life (t1/2) of GEN1057 | Predose and postdose at multiple timepoints up to end of treatment (approximately 4 months)
Clearance (CL) of GEN1057 From Plasma | Predose and postdose at multiple timepoints up to end of treatment (approximately 4 months)
Number of Participants with Anti-drug Antibodies (ADAs) to GEN1057 | Up to approximately 11 months
  Serum samples will be screened for ADAs binding to GEN1057 and the titer of confirmed positive samples will be reported.
Objective Response Rate (ORR) | Up to approximately 11 months
  The ORR is defined as the percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) based on response evaluation criteria in solid tumors (RECIST) version (v) 1.1 as assessed by the investigator.
Duration of Response (DOR) | Up to approximately 11 months
  DOR is defined as the time from the first documentation of response (CR or PR) to the date of progressive disease (PD) or death, whichever occurs earlier based on RECIST v1.1 as assessed by the investigator.
Time to Response (TTR) | Up to approximately 11 months
  TTR is defined as the time from Cycle 1 Day 1 (C1D1) to the first documentation of objective response (CR or PR) in participants achieving PR or CR based on RECIST v1.1 as assessed by the investigator.
Disease Control Rate (DCR) | Up to approximately 11 months
  DCR is defined as the percentage of participants with BOR of CR, PR, or stable disease (SD) based on RECIST v1.1 as assessed by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (5):
- United States (2):
  - SCRI Oncology Partners, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
- National Cancer Center, Tsukiji 5-1-1, Tokyo, Japan
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Start Madrid Centro Integral Oncologico Clara Campal CIOCC, Madrid

IPD SHARING:
Plan to Share IPD: No